CLINICAL TRIAL: NCT04778865
Title: Effect of Vitamin D Supplementation on Autoimmunity and Thyroid Function in Subjects With Hashimoto's Thyroiditis and Vitamin D Deficiency: Clinical Pilot Trial.
Brief Title: Effect of Treatment for Vitamin D Deficiency on Thyroid Function and Autoimmunity in Hashimoto's Thyroiditis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Claudia Vega Soto, Nutritionist, Universidad de Valparaiso
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 004/2020
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hashimoto Disease; Treatment Levothyroxine; Vitamin D Deficiency
Keywords: Hashimoto Disease; Vitamin D; Antithyroid antibodies; Thyroid stimulating hormone
MeSH Terms: conditions — Hashimoto Disease; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Patients will randomly receive the experimental condition or the active comparator for 3 months. After 3 months of washout, the groups will be crossed to receive the opposite treatment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D-correction (Experimental): Subjects will receive one capsule with 50.000 IU cholecalciferol weekly for 3 months.
  Interventions: Dietary Supplement: Vitamin D-correction
- Vitamin D-RDA (Active Comparator): Subjects will receive one capsule with 4.200 IU cholecalciferol weekly for 3 months.
  Interventions: Dietary Supplement: Vitamin D-RDA

INTERVENTIONS:
Dietary Supplement: Vitamin D-correction — Capsule with 50.000 UI cholecalciferol
  Arms: Vitamin D-correction
Dietary Supplement: Vitamin D-RDA — Capsule with 4.2000 UI cholecalciferol
  Arms: Vitamin D-RDA

SUMMARY:
The objective of this study is to evaluate the effect of vitamin D supplementation on thyroid autoimmunity, thyroid function, and other metabolic and clinical variables associated with the thyroid axis in patients with Hashimoto's thyroiditis and vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* women between 18-45 years old (pre-menopausal stage)
* men between 18-60 years old
* BMI between 18.5-34.9 kg/ m2
* medical diagnosis of Hashimoto's thyroiditis
* treatment with levothyroxine (LT4) with stable dose (from four months from the start of the intervention)
* positive antithyroid antibody (peroxidase and/or thyroglobulin)
* serum 25 (OH) D levels <20 ng / ml.

Exclusion Criteria:

* radioiodine, thyroidectomy, antithyroid treatment
* disease, condition or drug treatment that alters the immune system or hypothalamic-pituitary-thyroid axis or vitamin D metabolism.
* disorder of kidney, liver, or bone-metabolic function
* Graves disease, toxic nodular goiter, postpartum thyroiditis, coronary heart disease, epilepsy, cancer, Turner or Down syndrome, primary hyperparathyroidism
* vitamin D, calcium, complex B, omega-3 supplements
* pregnant or breastfeeding
* type 2 diabetes or dyslipidemia with drug treatment at unstable doses
* intense physical activity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline antithyroid antibodies at 3 months | Basal and final (after 3 months)
  Anti-thyroid peroxidase and anti-thyroglobulin antibodies (UI/mL)

SECONDARY OUTCOMES:
Change from baseline Thyroid stimulating hormone at 3 months | Basal and final (after 3 months)
  Serum Thyroid stimulating hormone (TSH) (uIU/mL)
Change from baseline Free thyroxine at 3 months | Basal and final (after 3 months)
  Serum Free thyroxine (FT4) (ng/dL)
Change from baseline Total triiodothyronine at 3 months | Basal and final (after 3 months)
  Serum Total triiodothyronine (T3) (ng/dL)
Change from baseline Lipid profile at 3 months | Basal and final (after 3 months)
  Lipid profile: It includes total cholesterol (mg/dl), high-density lipoprotein (HDL) (mg/dl), low-density lipoprotein (LDL) (mg/dl), very low-density lipoprotein (VLDL) (mg/dl), and triglycerides (mg/dl).
Change from baseline glycemia at 3 months | Basal and final (after 3 months)
  Fasting glycemia (mg/dl)
Change from baseline ThyPro-39 at 3 months | Basal and final (after 3 months)
  Questionnaire ThyPro-39 (Quality of Life Questionnaire for Patients with Thyroid Disease): ThyPRO-39 measures the severity of symptoms and overall health-related quality of life of patients with thyroid disease, self-reported during the previous 4 weeks through a questionnaire. Each item on the questionnaire is rated by a five-point Likert scale (not at all, a little, somewhat, quite a bit, very much/completely). ThyPRO-39 is made up of 39 items in13 scales: goiter symptoms; hyperthyroid symptoms; hypothyroid symptoms; eye symptoms; tiredness; cognitive complaints; anxiety; depressivity; emotional susceptibility; impaired social life; impaired daily life; cosmetic complaints/appearance; and overall quality of life (QoL)-impact scale.
Change from baseline SF-36 at 3 months | Basal and final (after 3 months)
  Questionnaire SF-36: The Short Form-36 Health Survey (SF-36) is a generic health-related quality of life (HRQL) questionnaires. The SF-36 Health Questionnaire is composed of 36 questions that assess health status through alternatives in items such as: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role and Mental health. Additionally, it includes an item on the change in general health status compared to the previous year.

OTHER OUTCOMES:
Change from baseline 25(OH)D at 3 months | Basal and final (after 3 months)
  25(OH)D (ng/mL)
Change from baseline Parathormone at 3 months | Basal and final (after 3 months)
  Parathormone (pg/mL)
Change from baseline calcium at 3 months | Basal and final (after 3 months)
  serum calcium (mg/dL)
Change from baseline phosphorus at 3 months | Basal and final (after 3 months)
  phosphorus (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Escuela de Nutrición. Facultad de Farmacia. Universidad de Valparaíso., Valparaíso, Chile